CLINICAL TRIAL: NCT06403943
Title: A Randomized, Controlled, Multicenter Clinical Study on the Efficacy and Safety of BaiDiZiYin Pill and ShenQiYiFei Pill as Adjunctive Treatments for Newly Diagnosed Pulmonary Tuberculosis Patients
Brief Title: Efficacy Safety BaiDiZiYin ShenQiYiFei Adjunctive Treatments Pulmonary Tuberculosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Shenyang Tenth People's Hospital (Other); Lanzhou Pulmonary Hospital (Unknown); Hebei Chest Hospital (Unknown); Anhui Chest Hospital (Other); Chongqing Public Health (Unknown); Chengdu Public Health Clinical Medical Center (Unknown); Guangzhou Chest Hospital. (Unknown); Third People's Court of Shenzhen (Unknown); Heilongjiang Provincial Institute of Infectious Disease Prevention and Control (Unknown); Wuhan tuberculosis Hospital (Unknown); Suzhou Fifth Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJCH-20240329
Record Dates: First submitted 2024-03-28; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Adjuvant; Treatment; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isoniazid; Rifampin; Ethambutol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): BaidiZiyin Wan and ShenqiYifei Wan are traditional Chinese medicines. Used as an adjuvant therapy for pulmonary tuberculosis. It is mainly used to improve the symptoms of tuberculosis (including fever, cough, expectoration, blood sputum or hemoptysis, anorexia, chest pain, emaciation, night sweats).
  Interventions: Drug: BaiDiZiYin Pill, ShenQiYiFei Pill; Drug: Anti tuberculosis chemotherapy
- Control group (Active Comparator): 2 months' intensive regimen of anti tuberculosis chemotherapy Recommended first-line anti tuberculosis regimen: 2HRZE
  Interventions: Drug: Anti tuberculosis chemotherapy

INTERVENTIONS:
Drug: BaiDiZiYin Pill, ShenQiYiFei Pill — Indications of BaidiZiyin Pill: Nourishing the lungs and kidneys, cooling blood and removing steam. Used as an adjunctive treatment for tuberculosis caused by lung and kidney deficiency and qi yin injury, including coughing, shortness of breath, dry cough with less phlegm, hot flashes and night sweats, cold and spontaneous sweating, hoarseness, palpitations, cold limbs, and emaciation.
  Indications of ShenqiYifei Pill: expectorant and cough relieving. It is suitable for patients with pulmonary tuberculosis and spleen diseases, as well as phlegm dampness retention. Symptoms include short breath, low sound, clear and thin phlegm, limited appetite, bloating and loose stools, pale complexion, fatigue and chest tightness, emaciation, and fear of cold and spontaneous sweating.
  Arms: Experimental group
Drug: Anti tuberculosis chemotherapy — 2 months' intensive regimen of anti tuberculosis chemotherapy Recommended first-line anti tuberculosis regimen: 2HRZE
  Other Names: 2 months Isoniazid, Rifampicin, Ethambutol, Pyrazinamide （2HRZE）

SUMMARY:
This study is designed to further strengthen the clinical application evidence of BaidiZiyin Pill and ShenqiYifei Pill in the treatment of tuberculosis. To be included in the initial treatment of pulmonary tuberculosis patients, on the basis of standardized Western medicine treatment, BaidiZiyin Pills and ShenqiYifei Pills will be used to evaluate the clinical efficacy and safety of their products.

1. Evaluate the improvement of symptoms in the adjuvant treatment of newly treated pulmonary tuberculosis with BaidiZiyin Pill and ShenqiYifei Pill.
2. Explore the sputum negative conversion time and sputum negative conversion rate of BaidiZiyin Pill and ShenqiYifei Pill as adjunctive treatments for newly treated pulmonary tuberculosis.
3. Explore the protective effects of BaidiZiyin Pill and ShenqiYifei Pill on adverse reactions caused by chemotherapy.

DETAILED DESCRIPTION:
1. Research drugs: Bai Di Zi Yin Wan and Shen Qi Yi Fei Wan.
2. Research objective: To evaluate the symptom improvement of Baidi Ziyin Pill and Shenqi Yifei Pill in the adjuvant treatment of newly treated pulmonary tuberculosis; Explore the sputum negative conversion time and sputum negative conversion rate of Baidi Ziyin Pill and Shenqi Yifei Pill as adjunctive treatments for newly treated pulmonary tuberculosis; Explore the protective effects of Baidi Ziyin Pill and Shenqi Yifei Pill on adverse reactions caused by chemotherapy.
3. Study design: A randomized, controlled, multicenter clinical study.
4. Clinical staging: re evaluation after listing.
5. Treatment plan:

Experimental group: Take Bai Di Zi Yin Wan in the morning, 45 pills per time; Take 45 pills of Shenqi Yifei Pill per time at night, combined with a first-line anti tuberculosis regimen of 2HRZE Control group: Antituberculosis chemotherapy Recommended frontline anti tuberculosis regimen: 2HRZE Isoniazid (0.3g), rifampicin (0.45g for weight 50kg and below, 0.6g for weight 50kg and above), pyrazinamide (1.5g), ethambutol (0.75g for weight 50kg and below, 1.0g for weight 50kg and above), once a day, for a course of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 65 years old, regardless of gender;
* 2. Meets the diagnostic criteria for Western medicine pulmonary tuberculosis (formulated in accordance with the health industry standard WS 288-2017 "Diagnosis of Pulmonary Tuberculosis" of the People's Republic of China [9])
* 3. Have not received anti tuberculosis treatment in the past, or have received HRZE anti tuberculosis treatment for less than 1 week as a first-line option
* 4. The subjects themselves have informed consent, voluntarily participate in this study, have good medication compliance, and have signed the subject's informed consent form.

Conforming to the diagnostic criteria for Qi and Yin deficiency syndrome in traditional Chinese medicine (in accordance with the industry standards of traditional Chinese medicine in the People's Republic of China - Traditional Chinese Medicine Internal Medicine - Diagnosis and Efficacy Criteria for Disease Symptoms ZY/T0011.1-94) Main symptoms: shortness of breath, fatigue, mental fatigue, weak pulse Secondary symptoms: hemoptysis, spontaneous sweating, night sweating, insufficient appetite, bloating, red and tender tongue, thin coating Diagnosis can be made by having two main symptoms and one secondary symptom.

Exclusion Criteria:

* 1. Patients who received similar traditional Chinese medicine treatment 4 weeks prior to enrollment;
* 2. Patients with drug-resistant and extensively drug-resistant pulmonary tuberculosis;
* 3. Known or suspected to have a history of allergies or serious adverse reactions to the investigational drug and its excipients, or allergic constitution.
* 4. Patients with drug sensitivity indicating the growth of non tuberculosis mycobacteria (more than twice) or clinically diagnosed with non tuberculosis mycobacterial disease or concomitant non tuberculosis mycobacterial disease;
* 5. For patients with recurrent pulmonary tuberculosis, those with bacterial negative pulmonary tuberculosis or those with initial bacterial positive pulmonary tuberculosis who have received anti tuberculosis treatment for more than one week;
* 6. Patients with combined autoimmune diseases, malignant tumors, severe hematological and hematopoietic system diseases, epilepsy, and psychiatric disorders;
* 7. Concomitant severe organic cardiovascular and cerebrovascular diseases (such as congestive heart failure, myocardial infarction, and acute stroke with NYHA heart function grading of III-IV);
* 8. Merge uncontrolled hypertension (blood pressure ≥ 160/100mmHg at enrollment);
* 9. diabetes with poor glycemic control;
* 10. Concomitant severe liver and kidney diseases, or abnormal liver and kidney function tests (ALT, AST ≥ 2.5 times the upper limit of normal, Scr>the upper limit of normal);
* 11. Patients with extrapulmonary tuberculosis such as lymph node tuberculosis, intestinal tuberculosis, bone tuberculosis, renal tuberculosis, epididymal tuberculosis, urogenital tuberculosis, nervous system tuberculosis, and tuberculous meningitis;
* 12. Concomitant with other lung diseases, such as lung tumors, cysts, abscesses, interstitial lung disease, silicosis, pneumoconiosis, etc
* 13. Pregnant and lactating women;
* 14. HIV patients; Syphilis antibody positive patients;
* 15. Individuals who have participated in other clinical trials within 15.1 months;
* 16. Those who suspect or have a history of alcohol or drug abuse or a tendency towards drug dependence;
* 17. The researchers believe that patients are not suitable for inclusion in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Improvement of symptoms | The Time Frame is 2 months. After 2 months, the following indicators are divided into: none (0 points); Light (1 point); Medium (2 points); Heavy (3 points).
  The change rate of symptoms and the overall clinical symptom score of pulmonary tuberculosis. The following indicators are divided into: none (0 points); Light (1 point); Medium (2 points); Heavy (3 points).
  Fatigue: None; Labor leads to fatigue; If you move, you will feel tired; Not moving is also lacking.
  Hemoptysis: None; Occasional hemoptysis or sputum with blood streaks; Occasional or minor hemoptysis; Frequent or moderate to massive hemoptysis.
  Cough: None; Intermittent coughing during the day does not affect work and life; Can persist in working despite coughing during the day or occasional coughing at night; Frequent coughing or working during the day and night can affect work and life.
  Phlegm: None; Cough 10-15ml of phlegm day and night; Cough 50-100ml of phlegm day and night; Coughing more than 100ml day and night.
  Chest pain: None; Mild chest pain; Chest pain is obvious but tolerable; Chest pain significantly affects respiratory cough.

CONTACTS AND LOCATIONS:
Overall Officials: WENJUAN NIE, DR, Study Director — Beijing Chest Hospital
Locations (1):
- Beijing Chest Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
1. Evaluate the improvement of symptoms in the adjuvant treatment of newly treated pulmonary tuberculosis with BaidiZiyin Pill and ShenqiYifei Pill.
  2. Explore the sputum negative conversion time and sputum negative conversion rate of BaidiZiyin Pill and ShenqiYifei Pill as adjunctive treatments for newly treated pulmonary tuberculosis.
  3. Explore the protective effects of BaidiZiyin Pill and ShenqiYifei Pill on adverse reactions caused by chemotherapy.
Supporting Information: Study Protocol
Time Frame: The data will become available in 2025 and for 5 years.
Access Criteria: Published on Journal.
URL: https://bmcinfectdis.biomedcentral.com